CLINICAL TRIAL: NCT07357571
Title: Multicenter Retrospective Study of Dual-mode Contrast-enhanced Ultrasound Predictive Model for Lymph Node Metastasis Burden in T1N0M0 Papillary Thyroid Carcinoma
Brief Title: Preoperative Prediction of Lymph Node Metastasis in T1N0M0 Papillary Thyroid Carcinoma by Using Contrast-enhanced Ultrasound
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jingliang Ruan, Associate Chief Physician, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2025-948-01
Record Dates: First submitted 2025-12-18; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Papillary Carcinoma; Contrast Enhanced Ultrasound
Keywords: thyroid papillary carcinoma; contrast enhanced ultrasound
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High Metastasis Burden Group: ≥5 involved lymph nodes or the maximum diameter of any involved lymph node ≥2 mm
- Low Metastasis Burden Group: <5 involved lymph nodes and the maximum diameter of all involved lymph nodes <2 mm.

SUMMARY:
Similarly, the burden of central lymph node metastasis affects the individualized management of patients with T1N0M0 papillary thyroid carcinoma (PTC): lymph node metastasis is a contraindication to thermal ablation; low-burden lymph node metastasis is suitable for lobectomy; and high-burden lymph node metastasis recommends total thyroidectomy. However, conventional preoperative imaging examinations have low efficacy in diagnosing central lymph node metastasis. This multicenter retrospective cross-sectional study enrolled 600 patients with T1N0M0 PTC who were admitted to our hospital from June 2018 to June 2025 and confirmed by postoperative pathology. Dynamic contrast-enhanced ultrasound (CEUS) images of the thyroid and lymph nodes before surgery were collected for all patients. Two senior ultrasound physicians unaware of the pathological results independently analyzed the images and extracted qualitative and quantitative CEUS features of lesions and suspicious lymph nodes. Taking postoperative pathological results as the gold standard, patients were divided into the high-burden metastasis group, low-burden metastasis group, and non-metastasis group. Univariate and multivariate Logistic regression analyses were used to screen independent predictors, construct a combined predictive model, and draw receiver operating characteristic (ROC) curves and decision curves to evaluate its diagnostic efficacy and clinical practicality. The primary outcome measure was the area under the curve (AUC), and the secondary outcome measures included sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and net benefit. This project is expected to achieve accurate preoperative prediction of the burden of central lymph node metastasis and realize precise and individualized treatment for patients with T1N0M0 PTC.

DETAILED DESCRIPTION:
Papillary thyroid carcinoma (PTC) is the most prevalent subtype of thyroid malignancy, accounting for approximately 80%-90% of all thyroid cancers globally. With the widespread application of high-resolution ultrasound in routine physical examinations, an increasing number of early-stage PTC cases, particularly those classified as T1N0M0 (tumor size ≤2 cm, no clinical evidence of lymph node metastasis, and no distant metastasis), are being detected. Despite the relatively favorable prognosis of T1N0M0 PTC, the presence and burden of central lymph node metastasis (CLNM) remain critical factors that directly guide individualized treatment strategies and long-term follow-up plans for patients.

Similarly, the burden of CLNM exerts a pivotal impact on the individualized management of T1N0M0 PTC patients, as distinct metastasis burdens correspond to significantly different therapeutic approaches. Specifically, lymph node metastasis of any burden serves as an absolute contraindication to thermal ablation, a minimally invasive treatment option increasingly used for low-risk PTC; patients with low-burden CLNM (defined as ≤3 positive central lymph nodes with no extracapsular extension) are typically suitable for thyroid lobectomy combined with central lymph node dissection, which balances tumor control and preservation of thyroid function; in contrast, high-burden CLNM (defined as >3 positive central lymph nodes or presence of extracapsular extension) recommends total thyroidectomy with comprehensive central lymph node dissection, followed by radioactive iodine therapy when necessary to reduce the risk of recurrence. However, conventional preoperative imaging examinations, including conventional ultrasound, computed tomography (CT), and magnetic resonance imaging (MRI), have inherent limitations in diagnosing CLNM and evaluating its burden. Conventional ultrasound relies primarily on morphological features (e.g., lymph node size, shape, cortical thickness) which lack sufficient specificity, while CT and MRI are associated with radiation exposure (for CT) or high cost (for MRI) and still demonstrate low sensitivity and specificity for detecting small or micrometastatic lymph nodes in the central compartment, leading to frequent misdiagnosis or underdiagnosis.

This limitation poses a clinical dilemma: inaccurate preoperative assessment of CLNM burden may result in overtreatment (e.g., unnecessary total thyroidectomy in patients with no or low-burden metastasis, leading to lifelong thyroid hormone replacement therapy) or undertreatment (e.g., lobectomy in patients with high-burden metastasis, increasing the risk of local recurrence and the need for reoperation). Therefore, there is an urgent clinical need for a non-invasive, accurate, and cost-effective imaging method to preoperatively evaluate the burden of CLNM in T1N0M0 PTC patients.

Dynamic contrast-enhanced ultrasound (CEUS) has emerged as a promising imaging technique in the field of thyroid and lymph node diagnostics. By intravenously injecting a microbubble contrast agent, CEUS can dynamically visualize the microvascular perfusion of target tissues in real time, providing qualitative (e.g., enhancement pattern, homogeneity, presence of perfusion defects) and quantitative (e.g., time to peak, peak intensity, wash-in rate, wash-out rate) parameters that reflect the pathological microenvironment of lesions. Compared with conventional imaging modalities, CEUS offers several advantages, including non-radiation exposure, real-time imaging, high spatial and temporal resolution, and the ability to assess microcirculation, which may enable more accurate identification of metastatic lymph nodes and evaluation of their burden.

To address the aforementioned clinical gap, this multicenter retrospective cross-sectional study was designed to explore the value of CEUS in preoperatively predicting the burden of CLNM in T1N0M0 PTC patients. The study enrolled 600 consecutive patients with T1N0M0 PTC who were admitted to three tertiary hospitals (the lead center and two collaborating centers) from June 2018 to June 2025 and confirmed by postoperative pathology. All patients met strict inclusion criteria: (1) histopathologically confirmed PTC after surgery; (2) preoperative tumor staging consistent with T1N0M0 based on clinical examination and conventional imaging; (3) no history of thyroid surgery, radioactive iodine therapy, or other malignant tumors; (4) availability of complete preoperative CEUS data of the thyroid and central compartment lymph nodes; and (5) no contraindications to contrast agent injection. Patients with incomplete clinical, imaging, or pathological data were excluded from the study.

Two senior ultrasound physicians with more than 10 years of experience in thyroid and lymph node imaging, who were completely blinded to the postoperative pathological results (including the presence and burden of CLNM), independently analyzed the stored CEUS images. They extracted a comprehensive set of qualitative and quantitative CEUS features. Qualitative features included: (1) enhancement pattern of the thyroid lesion (homogeneous vs. heterogeneous, hyperenhancement vs. hypoenhancement vs. isenhancement compared with surrounding normal thyroid tissue, presence of peripheral rim enhancement); (2) enhancement characteristics of suspicious lymph nodes (homogeneous vs. heterogeneous enhancement, presence of perfusion defects, cortical enhancement, medullary hilum disappearance); and (3) time sequence of enhancement (whether the lesion/lymph node enhances earlier or later than normal tissue). Quantitative features were measured using dedicated offline analysis software, including time to peak (TTP), peak intensity (PI), wash-in slope (WIS), wash-out rate (WOR), and area under the time-intensity curve (AUC-TIC) for both the thyroid lesion and suspicious lymph nodes.

Taking postoperative pathological results as the gold standard (the gold standard for CLNM diagnosis and burden assessment), patients were divided into three groups: (1) non-metastasis group: no positive central lymph nodes confirmed by pathology; (2) low-burden metastasis group: ≤3 positive central lymph nodes with no extracapsular extension; (3) high-burden metastasis group: >3 positive central lymph nodes or presence of extracapsular extension (extracapsular extension was defined as the infiltration of metastatic lymph node tissue beyond the lymph node capsule into adjacent soft tissues). Pathological examination was performed by two senior pathologists who were blinded to the CEUS results, and any discrepancies were resolved through consensus discussion.

Statistical analysis was performed using SPSS 26.0 and R 4.2.0 software. First, inter-observer agreement for qualitative and quantitative CEUS features was evaluated using the kappa coefficient (for qualitative features) and intraclass correlation coefficient (ICC) (for quantitative features), with kappa/ICC >0.75 indicating excellent agreement. Features with excellent inter-observer agreement were included in subsequent analyses. Then, univariate Logistic regression analysis was used to screen potential predictors of CLNM burden (i.e., comparing non-metastasis vs. metastasis, and low-burden vs. high-burden metastasis). Variables with a P value <0.1 in univariate analysis were included in multivariate Logistic regression analysis to identify independent predictors of CLNM burden. Based on the independent predictors, a combined predictive model was constructed, and the regression coefficient of each predictor was used to assign a weight to generate a risk score for CLNM burden.

To evaluate the diagnostic efficacy of the combined model, receiver operating characteristic (ROC) curves were drawn, and the area under the curve (AUC) was calculated as the primary outcome measure. The optimal cut-off value of the risk score was determined using the Youden index (sensitivity + specificity - 1). Secondary outcome measures included sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and accuracy, which were calculated based on the optimal cut-off value. Additionally, decision curve analysis (DCA) was performed to evaluate the clinical practicality of the model by quantifying the net benefit of using the model to guide clinical decision-making compared with the "treat all" or "treat none" strategies across different threshold probabilities.

This study is expected to achieve several key objectives: first, to identify the most valuable qualitative and quantitative CEUS features for predicting the burden of CLNM in T1N0M0 PTC; second, to construct a reliable combined predictive model based on these CEUS features that can accurately distinguish between non-metastasis, low-burden metastasis, and high-burden metastasis preoperatively; third, to validate the diagnostic efficacy and clinical applicability of the model through ROC and DCA analyses. Ultimately, this project aims to provide a non-invasive, accurate, and practical tool for preoperative assessment of CLNM burden in T1N0M0 PTC patients, thereby guiding clinicians to formulate more precise and individualized treatment plans, reducing the risk of overtreatment or undertreatment, improving patient prognosis, and optimizing the use of medical resources.

ELIGIBILITY:
Inclusion Criteria

1. Patients with preoperative assessment of T1N0M0 papillary thyroid carcinoma who underwent initial surgical treatment at the medical centers participating in this study between June 2018 and June 2025.
2. Definitive diagnosis of papillary thyroid carcinoma confirmed by postoperative histopathological examination.
3. Preoperative conventional ultrasound and contrast-enhanced ultrasound (CEUS) examination of the thyroid and/or suspicious central lymph nodes were performed, with complete imaging data of acceptable quality for analysis.
4. Surgical procedures included thyroidectomy (lobectomy or total thyroidectomy) combined with central lymph node dissection (prophylactic or therapeutic) to provide a definitive pathological gold standard for lymph nodes.
5. Complete clinical pathological data and imaging data were retrievable from the Hospital Information System (HIS).

Exclusion Criteria

1. Preoperative receipt of any anti-tumor treatment targeting the thyroid (e.g., radiotherapy, chemotherapy, targeted therapy, or ablation therapy).
2. Complication with other types of thyroid malignant tumors (e.g., medullary carcinoma, undifferentiated carcinoma, etc.).
3. History of neck surgery or radiotherapy that may affect the structure of cervical lymph nodes.
4. Complication with other systemic diseases that may affect CEUS perfusion characteristics or imaging evaluation (e.g., severe heart failure, liver cirrhosis, etc.).
5. Allergy to components of the ultrasound contrast agent.
6. Missing key clinical or imaging data, making complete analysis impossible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with T1N0M0 papillary thyroid carcinoma (PTC) who underwent initial surgical treatment and had preoperative evaluation confirmed as T1N0M0 at the medical centers participating in this study between June 2018 and June 2025.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Invasiveness | 2018-2025
  The burden of central lymph node metastasis. According to NCCN guidelines, The burden of central lymph node metastas is categorized as "high" (≥5 involved nodes or any metastatic focus ≥2 mm), "low" (<5 involved nodes and all metastatic foci <2 mm), and "none" (no central lymph node metastasis).

CONTACTS AND LOCATIONS:
Overall Officials: Jingliang Ruan, Doctoral Degree, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (2):
- China (2):
  - Sun Yat-sen Memorial Hospital, Guangdong, Guangzhou
  - No. 33 Yingfeng Road, Haizhu District, Guangzhou City, Guangdong Province, Sun Yat-sen Memorial Hospital, Guangzhou, Guangzhou

IPD SHARING:
Plan to Share IPD: Yes
1. Preoperative dual-modality ultrasound files/reports (conventional/CEUS features of lesions/central lymph nodes);
  2. Clinical baseline data (age, gender, pathology subtype, TNM stage, thyroid function);
  3. Postoperative pathology data (metastatic central lymph node count, focus diameter). All data are anonymized (no personal info) to protect privacy. Eligible researchers (with ethics approval for thyroid cancer studies) may apply via the study's encrypted platform 12 months post-study completion. IPD is for non-commercial academic use only.
Supporting Information: Study Protocol
Time Frame: 2025-2026
Access Criteria: Eligible academic researchers (with ethics committee approval for thyroid cancer imaging-related studies) may access the de-identified IPD (including dual-modality ultrasound data, clinical baseline records, and postoperative pathology results of thyroid carcinoma patients). To request access, researchers need to submit a formal application to the study leading team (via email) detailing their research purpose; after review and approval, they will receive access credentials for the study's encrypted secure data-sharing platform.

REFERENCES:
- [Background] Riley RD, Ensor J, Snell KIE, Harrell FE Jr, Martin GP, Reitsma JB, Moons KGM, Collins G, van Smeden M. Calculating the sample size required for developing a clinical prediction model. BMJ. 2020 Mar 18;368:m441. doi: 10.1136/bmj.m441. No abstract available. PMID 32188600
- [Background] Riley RD, Collins GS, Ensor J, Archer L, Booth S, Mozumder SI, Rutherford MJ, van Smeden M, Lambert PC, Snell KIE. Minimum sample size calculations for external validation of a clinical prediction model with a time-to-event outcome. Stat Med. 2022 Mar 30;41(7):1280-1295. doi: 10.1002/sim.9275. Epub 2021 Dec 16. PMID 34915593
- [Background] Luo ZY, Hong YR, Yan CX, Wang Y, Ye Q, Huang P. Utility of quantitative contrast-enhanced ultrasound for the prediction of lymph node metastasis in patients with papillary thyroid carcinoma. Clin Hemorheol Microcirc. 2022;80(1):37-48. doi: 10.3233/CH-200909. PMID 33252064
- [Background] Yu Y, Shi LL, Zhang HW, Wang Q. Performance of contrast-enhanced ultrasound for lymph node metastasis in papillary thyroid carcinoma: a meta-analysis. Endocr Connect. 2023 Jan 19;12(2):e220341. doi: 10.1530/EC-22-0341. Print 2023 Feb 1. PMID 36524799
- [Background] Li QL, Ma T, Wang ZJ, Huang L, Liu W, Chen M, Sang T, Ren XG, Tong J, Cao CL, Dong J, Li J. The value of contrast-enhanced ultrasound for the diagnosis of metastatic cervical lymph nodes of papillary thyroid carcinoma: A systematic review and meta-analysis. J Clin Ultrasound. 2022 Jan;50(1):60-69. doi: 10.1002/jcu.23073. Epub 2021 Oct 8. PMID 34625988
- [Background] Yang Z, Wang X, Tao T, Zou J, Qiu Z, Wang L, Du H, Chen N, Yin X. Diagnostic value of contrast-enhanced ultrasonography in the preoperative evaluation of lymph node metastasis in papillary thyroid carcinoma: a single-center retrospective study. BMC Surg. 2023 Oct 24;23(1):325. doi: 10.1186/s12893-023-02199-w. PMID 37875825
- [Background] Chen L, Chen L, Liang Z, Shao Y, Sun X, Liu J. Value of Contrast-Enhanced Ultrasound in the Preoperative Evaluation of Papillary Thyroid Carcinoma Invasiveness. Front Oncol. 2022 Jan 14;11:795302. doi: 10.3389/fonc.2021.795302. eCollection 2021. PMID 35096595
- [Background] Hong YR, Luo ZY, Mo GQ, Wang P, Ye Q, Huang PT. Role of Contrast-Enhanced Ultrasound in the Pre-operative Diagnosis of Cervical Lymph Node Metastasis in Patients with Papillary Thyroid Carcinoma. Ultrasound Med Biol. 2017 Nov;43(11):2567-2575. doi: 10.1016/j.ultrasmedbio.2017.07.010. Epub 2017 Aug 12. PMID 28807450
- [Background] Yang J, Zhang F, Qiao Y. Diagnostic accuracy of ultrasound, CT and their combination in detecting cervical lymph node metastasis in patients with papillary thyroid cancer: a systematic review and meta-analysis. BMJ Open. 2022 Jul 4;12(7):e051568. doi: 10.1136/bmjopen-2021-051568. PMID 35788082
- [Background] Zhao F, Wang P, Yu C, Song X, Wang H, Fang J, Zhu C, Li Y. A LASSO-based model to predict central lymph node metastasis in preoperative patients with cN0 papillary thyroid cancer. Front Oncol. 2023 Jan 25;13:1034047. doi: 10.3389/fonc.2023.1034047. eCollection 2023. PMID 36761950
- [Background] Zheng WH, Li C, Sun RH, Shui CY, Wang X, He TQ, Cai YC, Ning YD, Jiang J, Qin G, Zhou YQ, Liu W. [Advances in the research of central lymph node dissection for cN0 thyroid papillary carcinoma]. Zhonghua Er Bi Yan Hou Tou Jing Wai Ke Za Zhi. 2020 Aug 7;55(8):799-803. doi: 10.3760/cma.j.cn115330-20200411-00289. Chinese. PMID 32791784